CLINICAL TRIAL: NCT02522936
Title: Use of Biotene Moisturizing Mouth Spray for Xerostomia Associated With Oral Oxybutynin Use
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to lack of funding and necessary personnel we determined that the study could not be done.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Begum Ozel, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-14-00800
Record Dates: First submitted 2015-08-12; First posted 2015-08-13 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Overactive Bladder; Xerostomia; Compliance
MeSH Terms: conditions — Urinary Bladder, Overactive; Xerostomia; Patient Compliance | interventions — Biotene

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biotene (Experimental): Participants will be given Biotene oral spray to use as needed when taking oxybutynin.
  Interventions: Drug: Biotene oral spray
- Routine care (No Intervention): Participants will be given routine care.

INTERVENTIONS:
Drug: Biotene oral spray — Biotene oral spray will be provided to participants.
  Other Names: Biotene; Mouth spray
  Arms: Biotene

SUMMARY:
This is a randomized placebo controlled trial of the use of Biotene versus no treatment in women receiving oral oxybutynin for overactive bladder. The primary outcome will be rate of discontinuation of oxybutynin at 6 month.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a common condition affecting roughly 20% of women. Anticholinergic medications are the main treatment modality for women with OAB; however, treatment is hampered by high rates of dry mouth which limit tolerability. Discontinuation rates for anticholinergic medications for dry mouth have been reported to be as high as 71% at 6 months. Biotène(TM) Moisturizing Mouth Spray is used for xerostomia due to various etiologies in adults.

The purpose of our study is to determine the rate of discontinuation of oral oxybutynin therapy for overactive bladder in women using Biotène(TM) Moisturizing Mouth Spray versus no additional treatment. This is a randomized open label trial. Participants will be randomized to moisturizing mouth spray versus no additional treatment. Urinary symptoms, xerostomia symptoms, and compliance with oral oxybutynin will be compared between groups. Our primary outcome is rate of discontinuation of oral oxybutynin at 6 months.

Assuming a baseline discontinuation rate of 70% at 6 months, and assuming 80% power and α = 0.05 for a two-sided test, we will require 42 subjects in each group to detect a difference of 30% in cure rate between the two groups. Assuming followup of 75%, 60 subjects in each group will be recruited.

Participants within groups will be compared with respect to differences in baseline demographics, questionnaire scores and compliance with oxybutynin using a Chi Square test for categorical variable, a T test for normally distributed continuous variables or a Mann Whitney U test for non-normally distributed or ordinal variables.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Able to give informed consent
* Women diagnosed with overactive bladder or urgency incontinence who are being started on oral oxybutynin.

Exclusion Criteria:

* Any allergy to Biotène® Moisturizing Mouth Spray or its components
* Any contraindication to oxybutynin, including urinary retention (PVR > 100ml), gastric retention and other severe decreased gastrointestinal motility conditions, uncontrolled narrow-angle glaucoma and in patients who are at risk for these conditions, and patients who have demonstrated hypersensitivity to the drug substance or other components of the product.
* Using ocular anti-cholinergic agents, treatment for dry mouth or oral anti-muscarinics in the preceding 3 months.
* Prior history of head/neck surgery or radiation (excluding thyroid surgery).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Discontinuation rate of oxybutynin at 6 month by patient report | 6 months

SECONDARY OUTCOMES:
Discontinuation rate of oxybutynin at 6 months based on pill count | 6 months
Discontinuation rate of oxybutynin at 3 months as measured by patient report | 3 months
Discontinuation rate of oxybutynin at 3 months as measured by pill count | 3 months
Symptoms of dry mouth as measured by global xerostomia question | 3 months
Number of daily voids as measured by voiding diary | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dancz, Study Chair — University of Southern California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Versi E, Appell R, Mobley D, Patton W, Saltzstein D. Dry mouth with conventional and controlled-release oxybutynin in urinary incontinence. The Ditropan XL Study Group. Obstet Gynecol. 2000 May;95(5):718-21. doi: 10.1016/s0029-7844(99)00661-4. PMID 10775736
- [Result] Epstein JB, Emerton S, Le ND, Stevenson-Moore P. A double-blind crossover trial of Oral Balance gel and Biotene toothpaste versus placebo in patients with xerostomia following radiation therapy. Oral Oncol. 1999 Mar;35(2):132-7. doi: 10.1016/s1368-8375(98)00109-2. PMID 10435146
- [Result] Nelken RS, Ozel BZ, Leegant AR, Felix JC, Mishell DR Jr. Randomized trial of estradiol vaginal ring versus oral oxybutynin for the treatment of overactive bladder. Menopause. 2011 Sep;18(9):962-6. doi: 10.1097/gme.0b013e3182104977. PMID 21532512
- [Result] Matear DW, Barbaro J. Effectiveness of saliva substitute products in the treatment of dry mouth in the elderly: a pilot study. J R Soc Promot Health. 2005 Jan;125(1):35-41. doi: 10.1177/146642400512500113. PMID 15712851
- [Result] Thomson WM, van der Putten GJ, de Baat C, Ikebe K, Matsuda K, Enoki K, Hopcraft MS, Ling GY. Shortening the xerostomia inventory. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Sep;112(3):322-7. doi: 10.1016/j.tripleo.2011.03.024. Epub 2011 Jul 16. PMID 21684773